CLINICAL TRIAL: NCT02567695
Title: A Phase 1, Single-Dose, Open-Label, Randomized, Two-Period Crossover Study to Evaluate the Relative Bioavailability of GBT440 300 mg Administered as Capsule Formulations in Healthy Subjects
Brief Title: A Single-Dose Relative Bioavailability Study Of GBT440 300 mg Capsules in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Blood Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GBT440-004
Record Dates: First submitted 2015-09-30; First posted 2015-10-05 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2015-09

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence 1 (Experimental): Treatment A with one 300 mg capsule (high-strength) of GBT440 administered in a fasted state (test) in dosing Period 1 followed by Treatment B with 300 mg (3 × 100 mg) capsules (low-strength) of GBT440 administered in a fasted state (reference) in dosing Period 2.
  Interventions: Drug: GBT440
- Treatment Sequence 2 (Experimental): Treatment B with 300 mg (3 × 100 mg) capsules (low-strength) of GBT440 administered in a fasted state (reference) in dosing Period 1 followed by Treatment A with one 300 mg capsule (high-strength) of GBT440 administered in a fasted state (test) in dosing Period 2.
  Interventions: Drug: GBT440

INTERVENTIONS:
Drug: GBT440 — Test: GBT440 300 mg capsule (high-strength) Reference: GBT440 100 mg capsule (low-strength)

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of a single 300 mg dose of GBT440 administered as a high strength (1 × 300 mg) capsule versus a low strength (3 × 100 mg) capsule formulation in healthy fasted subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a female of non-childbearing potential or male, who is healthy, nonsmoking, and 18 to 60 years old, inclusive, at screening
* Male subjects agree to use contraception
* Willing and able to give written informed consent

Exclusion Criteria:

* Evidence or history of clinically significant metabolic, allergic, dermatological, hepatic, renal,hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* History of hypersensitivity or allergy to drugs, foods, or other substances
* History or presence of abnormal electrocardiogram or hypertension
* History of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or any history of drug abuse or addiction within 1 year of screening
* Participated in another clinical trial of an investigational drug within 30 days (or 5 half-lives of the investigational drug, whichever is longer) prior to Screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum observed concentration (Cmax) of GBT440 in whole blood | predose, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose, and Day 12, Day 20, and Day 28 for each period
Pharmacokinetics (PK): Area under the concentration-time curve (AUC) from time 0 to the time of the last quantifiable concentration (AUCt) of GBT440 in whole blood | predose, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose, and Day 12, Day 20, and Day 28 for each period
Pharmacokinetics (PK): AUC from time 0 extrapolated to infinity (AUCinf) of GBT440 in whole blood | predose, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose, and Day 12, Day 20, and Day 28 for each period

SECONDARY OUTCOMES:
Pharmacokinetics (PK): The time that Cmax was observed (tmax) of GBT440 in whole blood | predose, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose, and Day 12, Day 20, and Day 28 for each period
Pharmacokinetics (PK): Terminal elimination half-life (t½) of GBT440 in whole blood | predose, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose, and Day 12, Day 20, and Day 28 for each period
Pharmacokinetics (PK): Apparent oral clearance (CL/F) of GBT440 in whole blood | predose, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose, and Day 12, Day 20, and Day 28 for each period
Pharmacokinetics (PK): Apparent volume of distribution during the terminal phase (Vz/F) of GBT440 in whole blood | predose, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72, and 96 hours postdose, and Day 12, Day 20, and Day 28 for each period

OTHER OUTCOMES:
Treatment-emergent adverse events (TEAEs) and serious adverse events | Baseline to Period 2 Day 28
Changes in clinical laboratory results | Baseline to Period 2 Day 28
Changes in physical examination findings | Baseline to Period 2 Day 28
Changes in vital signs | Baseline to Period 2 Day 28
Changes in electrocardiograms (ECGs) | Baseline to Period 2 Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Carla Washington, PhD, Study Director — Global Blood Therapeutics
Locations (1):
- ICON Early Phase Services, LLC Clinical Research Unit, San Antonio, Texas, United States